CLINICAL TRIAL: NCT00437099
Title: Efficacy of Omega-3 Fatty Acids on Borderline Personality Disorder: a Randomized, Double Blind Clinical Trial.
Brief Title: Efficacy of Omega-3 Fatty Acids on Borderline Personality Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Miguel Casas Brugué, s
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TLP-OMEGA 3
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Borderline Personality Disorder.
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): subjects with BPD receiving Omacor 1.680 mg/d
  Interventions: Drug: Omacor®
- 2 (Experimental): BPD patients randomized to Omacor 3.360 mg/d
  Interventions: Drug: Omacor®
- 3 (Placebo Comparator): patients with BPD randomized to Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omacor® — arm 1: Omacor 1680 Arm 2: Omacor 3360
  Arms: 1; 2
Drug: Placebo — Placebo
  Arms: 3

SUMMARY:
Borderline Personality Disorder (BDP) is a serious mental disorder that affects about 1-2% of the general population, and it is characterized by severe psychosocial impairment and a high mortality rate due to suicide. Currently, the most effective treatments for BPD are psychotherapy (cognitive behavior therapy - CBT -) and pharmacotherapy (often as an important adjunctive role, especially for diminution of symptoms such as affective instability, impulsivity, psychotic-like symptoms and self-destructive behavior). Nevertheless, although several drugs are used in these patients, these drugs induce an improvement of some symptoms but do not cause the remission of BPD. Thus, identification of novel treatments is needed.

The objective of this study is to examine the efficacy of Omacor® ( a mixture of omega-3-acid ethyl esters: eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) ) for BDP patients receiving CBT. Patients with BDP will be randomly allocated to the three arms of the study: 1- CBT+placebo, 2- CBT+Omacor 1680 mg/d, 3- CBT+Omacor 3360 mg/d. Follow up will last for 12 weeks. Assessment of affective symptoms, impulsivity and aggressivity will be carried out at baseline and at 2, 4, 6, 8, 10 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Meet DSM-IV criteria for BPD assessed by the Structured Clinical Interview for DSM-IV Personality Disorders (SCID-II).
2. Clinical Global Impression of Severity for BDP > 3.
3. Age between 18 and 65 years.
4. Be able to give informed consent for participation.
5. Place of residency compatible with the assistance to the center.
6. If woman, use of effective contraception.

Exclusion Criteria:

1. Have a serious medical illness.
2. History of omacor® allergy.
3. Current diagnostic unipolar depression, bipolar disorder type I, Obsessive-Compulsive Disorder, schizophrenia and other psychotic disorders.
4. DIB-R > 8.
5. Suicidal thinking that requires hospital admission.
6. Meet DSM-IV criteria for alcohol, benzodiazepine, opioid or psychostimulant dependence in the six months prior to trial entry.
7. Transaminase elevation within three times the upper limits of normality.
8. Treatment with stable doses of antidepressants or mood stabilizers for less than six weeks.
9. Treatment with stable doses of antipsychotics for more than 1 week in the last three months.
10. Have received electroconvulsive therapy for the six months prior to trial entry.
11. Have received DBT in the last 12 months prior to trial entry.
12. Are pregnant or nursing.
13. Have participated in any other investigational study in the last 6 months prior to trial entry.
14. Current treatment or expectation to start any treatment with drugs that may interact with the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Affective symptoms measured with the Hamilton Depression Scale (Ham-D) and the Young Mania Rating Scale (YMRS). | weeks: 0, 2, 4, 6, 8, 10, 12
Impulsivity and aggressivity measured with the Time Paradigsm and the the Point Subtraction Aggression Paradigm. | 0, 6, 12

SECONDARY OUTCOMES:
Impulsivity assessed by means of Barratt Impulsivity Scale-11 (BIS-11) | Weeks 0, 2, 4, 6, 8, 10, 12
Anger assessed by means of the State-Trait Anger Expression Inventory 2 (STAXI-2) | Weeks 0, 2, 4, 6, 8, 10, 12
anxiety assessed by means of the State-Trait Anxiety Inventory (STAI-E) | weeks: 0, 6, 12
Brief Psychiatric Rating Scale (BPRS) | Weeks: 0, 6, 12
Global Activity Scale (EEAG) | Weeks: 0, 6, 12
Consumption of addictive substances with urine and breath drug testings and self-reports. | Every week throghout the study
Social Adaptation Self-evaluation Scale (SASS) | Weeks: 0, 6, 12
Number of suicidal and parasuicidal episodes. | Every week throughout the study
Number of visits to a psychiatric emergency service. | Every week throughout the study
Plasmatic BDNF. | Weeks 0, 12
Adverse events. | Every week throughout the study
Clinical impression assessed by means ICG | weeks: 0, 2, 4, 6, 8, 10, 12
Adverse events | at each study visit
immediate memory assessed by means of the Immediate Memory Task | Weeks 0, 6, 12
Impulsivity assessed by means the two choice delayed reward test | weeks: 0, 6, 12

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Casas, MD., Prof., Principal Investigator — Hospital Universitari Vall d'Hebron Barcelona, Catalonia, Spain
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Stoffers-Winterling JM, Storebo OJ, Pereira Ribeiro J, Kongerslev MT, Vollm BA, Mattivi JT, Faltinsen E, Todorovac A, Jorgensen MS, Callesen HE, Sales CP, Schaug JP, Simonsen E, Lieb K. Pharmacological interventions for people with borderline personality disorder. Cochrane Database Syst Rev. 2022 Nov 14;11(11):CD012956. doi: 10.1002/14651858.CD012956.pub2. PMID 36375174